CLINICAL TRIAL: NCT02779751
Title: A Phase 1b Study of Abemaciclib in Combination With Pembrolizumab for Patients With Stage IV Non-Small Cell Lung Cancer or Hormone Receptor Positive, HER2 Negative Breast Cancer
Brief Title: A Study of Abemaciclib (LY2835219) in Participants With Non-Small Cell Lung Cancer or Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16177; I3Y-MC-JPCE (Other: Eli Lilly and Company); 2015-005156-94 (EudraCT Number); KEYNOTE 287 (Other: Merck)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2016-05-19; First posted 2016-05-20 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer; Breast Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Breast Neoplasms | interventions — abemaciclib; pembrolizumab; Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- NSCLC KRAS mt, PD-L1+ (Experimental): Abemaciclib given orally every 12 hours (Q12H) on days 1 to 21 of each 21 day cycle in combination with pembrolizumab given intravenously (IV) on day 1 of each 21 day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Abemaciclib; Drug: Pembrolizumab
- NSCLC Squamous (Experimental): Abemaciclib given orally Q12H on days 1 to 21 of each 21 day cycle in combination with pembrolizumab given IV on day 1 of each 21 day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Abemaciclib; Drug: Pembrolizumab
- HR+, HER2- Metastatic Breast Cancer (Experimental): Abemaciclib given orally Q12H on days 1 to 21 of each 21 day cycle in combination with pembrolizumab given IV on day 1 of each 21 day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Abemaciclib; Drug: Pembrolizumab
- HR+, HER2- Locally Advanced or Metastatic Breast Cancer (Experimental): Abemaciclib given orally Q12H on days 1 to 21 of each 21 day cycle in combination with pembrolizumab given IV on day 1 of each 21 day cycle and anastrozole given orally Q24H on days 1 to 21 of each 21 day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Abemaciclib; Drug: Pembrolizumab; Drug: Anastrozole

INTERVENTIONS:
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
Drug: Pembrolizumab — Administered IV
Drug: Anastrozole — Administered orally
  Arms: HR+, HER2- Locally Advanced or Metastatic Breast Cancer

SUMMARY:
The main purpose of this study is to evaluate the safety and efficacy of abemaciclib in combination with pembrolizumab in participants with advanced non-small cell lung cancer (NSCLC) or hormone receptor positive (HR+), human epidermal growth factor receptor negative (HER2-) breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have a Stage IV diagnosis of 1 of the following: Part A: NSCLC (Kirsten rat sarcoma mutant [KRAS mt], PD-L1+); Part B: NSCLC (squamous histology); Part C: metastatic breast cancer (HR+, HER2-); or Part D: locally advanced or metastatic breast cancer (HR+, HER2-)

  * Part A: must be chemotherapy naïve for metastatic NSCLC
  * Part B: must have received at least 1 prior therapy containing platinum-based chemotherapy for advanced/metastatic NSCLC
  * Part C: must have previously received prior treatment with at least 1 but no more than 2 chemotherapy regimens in the metastatic setting
  * Part D: cannot have received endocrine therapy or chemotherapy as treatment in the locoregionally recurrent or metastatic breast cancer disease setting. Note: Participants may be enrolled if they received prior (neo)adjuvant chemotherapy or endocrine therapy for localized disease.
* Are amenable to provide tumor tissue prior to treatment and provide tumor tissue after treatment initiation (both mandatory).
* Have presence of measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
* Have a performance status (PS) ≤1 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Have discontinued all previous treatments for cancer and recovered from the acute effects of therapy.
* Have an estimated life expectancy of ≥12 weeks.
* For Part D: Have postmenopausal status due to surgical/natural menopause or chemical ovarian suppression (initiated 28 days prior to Day 1 of Cycle 1) with a gonadotropin-releasing hormone (GnRH) agonist such as goserelin or radiation-induced ovarian suppression.

Exclusion Criteria:

* Have a personal history of any of the following conditions: syncope of either unexplained or cardiovascular etiology, ventricular arrhythmia (including but not limited to ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest. Exception: subjects with controlled atrial fibrillation for >30 days prior to study treatment are eligible.
* Have central nervous system (CNS) metastasis with development of associated neurological changes 14 days prior to receiving study drug.
* Have corrected QT interval of >470 milliseconds on screening electrocardiogram (ECG).
* Have history of interstitial lung disease or pneumonitis.
* Have history of or active autoimmune disease, or other syndrome that requires systemic steroids or autoimmune agents for the past 2 years.
* Have received a live vaccination within 30 days of study start.
* Have received prior treatment with an anti PD-1, anti-programmed death ligand 1 (PD-L1), or anti cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) agent.
* For Part D Only:

  * Have initiated bisphosphonates or approved RANK ligand (RANK-L) targeted agents (for example, denosumab) <7 days prior to Cycle 1 Day 1.
  * Are currently receiving or have previously received endocrine therapy for locoregionally recurrent or metastatic breast cancer. Note: A participant may be enrolled if she received prior (neo)adjuvant endocrine therapy (including, but not limited to anti-estrogens or aromatase inhibitors) for localized disease.
  * Are currently receiving or have previously received chemotherapy for locoregionally recurrent or metastatic breast cancer. Note: Participants may be enrolled if they received prior (neo)adjuvant chemotherapy for localized disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-11-14 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) | Baseline through Study Treatment Completion (Approximately 6 Months)
Number of Participants with Non-Serious Adverse Event(s) | Baseline through Study Treatment Completion (Approximately 6 Months)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per RECIST v1.1: Percentage of Participants With a Complete or Partial Response | Baseline to Measured Progressive Disease or Start of New Anti-Cancer Therapy (Approximately 6 Months)
Disease Control Rate (DCR) per RECIST v1.1: Percentage of Participants With a Best Overall Response of Complete Response, Partial Response, and Stable Disease | Baseline to Measured Progressive Disease or Start of New Anti-Cancer Therapy (Approximately 6 Months)
Duration of Response (DoR) per RECIST v1.1 | Date of Complete Response or Partial Response to Date of Objective Disease Progression or Death Due to Any Cause (Approximately 12 Months)
Progression Free Survival (PFS) per RECIST v1.1 | Baseline to Measured Progressive Disease or Death (Approximately 10 Months)
Overall Survival (OS) | Baseline to Date of Death Due to Any Cause (Approximately 18 Months)
Pharmacokinetics (PK): Mean Steady State Exposure of Abemaciclib in Combination with Pembrolizumab with or without Anastrozole | Predose Cycle One Day One through Predose Cycle Eight Day One (21 Day Cycles)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (24):
- United States (7):
  - Highlands Oncology Group - Duplicate 2, Springdale, Arkansas
  - Univ of California San Francisco, San Francisco, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute, Farmington Hills, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
- Belgium (2):
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire Sart Tilman, Liège
- France (3):
  - Centre Oscar Lambret, Lille, Hauts-de-France
  - Hôpital Arnaud de Villeneuve - CHU Montpellier, Montpellier, Hérault
  - Hopital Larrey, Toulouse
- Italy (2):
  - Istituto Scientifico Romagnolo - Studio e la Cura dei Tumori, Meldola, Forli
  - IRCCS Ospedale San Raffaele, Milan
- Spain (4):
  - Hospital Nuestra Senora de Sonsoles, Ávila
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Madrid Norte Sanchinarro, Madrid
- Taiwan (4):
  - Tri-Service General Hospital, Neihu Taipei
  - Taipei Medical University- Shuang Ho Hospital, New Taipei City
  - Chi Mei Hospital - Liouying Branch, Tainan
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (2):
  - Istanbul Universitesi-Cerrahpasa Cerrahpasa Tip Fakultesi Yerleskesi, Istanbul
  - Ege Universitesi Hastanesi, Izmir

REFERENCES:
- [Derived] Pujol JL, Vansteenkiste J, Paz-Ares Rodriguez L, Gregorc V, Mazieres J, Awad M, Janne PA, Chisamore M, Hossain AM, Chen Y, Beck JT. Abemaciclib in Combination With Pembrolizumab for Stage IV KRAS-Mutant or Squamous NSCLC: A Phase 1b Study. JTO Clin Res Rep. 2021 Sep 25;2(11):100234. doi: 10.1016/j.jtocrr.2021.100234. eCollection 2021 Nov. PMID 34746886
- See also: A Study of Abemaciclib (LY2835219) in Participants With Non-Small Cell Lung Cancer or Breast Cancer — https://trials.lillytrialguide.com/en-US/trial/7MTCU0kNXyEgCUKm0oQgIY